CLINICAL TRIAL: NCT01504217
Title: Analysis of Muscle Strength and Control of Center of Mass Acceleration Mechanism to Predict Balance Ability and Fall Risks in Elderly
Brief Title: Control of Center of Mass to Predict Balance Ability and Fall Risks in Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200912073R
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Healthy older people over 65 years old

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Falling among older adults is a major public health concern. In fact, falls are the leading cause of accidental death in older adults both in Taiwan and in the United States. In order to provide effective preventative strategies, the investigators must understand the mechanisms that cause older adults to fall. Thus, the investigators research aim for three objectives: (1) using biomechanical model to identify the deficits in neuromuscular control for older adults (2) to apply research findings to the development of new clinical methods for assessing and recovering balance control in older adults, and (3) to predict fall risks in 1-2 year for older adults from the research findings.

ELIGIBILITY:
Inclusion Criteria:

1. can stand for 5 minutes without support
2. with normal or corrected to normal vision
3. age between 20-35 years old for young adults group, and 65-80 years old for older adults group
4. had fall history in the past 3 years for the older adults group.

Exclusion Criteria:

1. pregnant women
2. with cancer diagnosis
3. with sensory-motor deficits
4. with osteoporosis for older adults group (T-score below -2.5)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, PT, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- School & Graduate Institute of Physical Therapy College of Medicine, National Taiwan University, Taipei, Taiwan